CLINICAL TRIAL: NCT00549614
Title: Effect of 4 Weeks Treatment With Acipimox on Left Ventricular Function, Work Capacity, Insulin Sensitivity and Substrate Metabolism in Patients With Chronic Heart Failure
Brief Title: Effect of 4 Weeks Treatment With Acipimox in Patients With Chronic Heart Failure
Acronym: ACME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Cand. Med. Mads Halbirk, Department of Cardiology, Aarhus Universityhospital, Skejby
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20061218
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: acipimox
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acipimox — capsule, 250 mg, 4 times daily for 28 days
  Arms: 1
Drug: placebo — capsule, 250 mg, 4 times daily for 28 days
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate whether metabolic modulation improves left ventricular function, work capacity, insulin sensitivity and modifies substrate metabolism in chronic heart failure

ELIGIBILITY:
Inclusion Criteria:

* EF<40 %
* IHD
* NYHA-class II-III.

Exclusion Criteria:

* pregnancy
* severe renal failure
* new brady- or tachyArrhythmia
* Severe stenotic valvular disease
* myocardial infarction within last 6 weeks
* insulin treated diabetes mellitus
* peptic ulcer
* pregnancy or lactating women
* allergy towards tested medicine

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
left ventricular ejection Fraction | 4 weeks
exercise capacity | 4 weeks
muscular metabolism | 4 weeks

SECONDARY OUTCOMES:
regional left ventricular function | 4 weeks
insulin resistance | 4 weeks
full body metabolism | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mads Halbirk, Principal Investigator — B-research, Aarhus Universityhospital, skejby
Locations (1):
- Department of Cardiology, Aarhus Universityhospital, Skejby, Aarhus N, Denmark